CLINICAL TRIAL: NCT01386749
Title: The Efficacy of Low-Magnitude, High Frequency Vibration Treatment on Accelerating the Healing of Femoral Shaft Fracture - A Prospective Randomized Controlled Clinical Trial
Brief Title: Effect of Low-Magnitude, High Frequency Vibration Treatment on Femoral Shaft Fracture Healing
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kwok-Sui Leung, Chair Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 470410
Record Dates: First submitted 2011-06-22; First posted 2011-07-01 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Fracture, Closed, Comminuted, Healing
Keywords: Vibration treatment; Fracture healing; Muscular function
MeSH Terms: conditions — Fractures, Bone; Fractures, Comminuted

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Treatment (Experimental): receive 6 months LMHFV
  Interventions: Procedure: vibration platform provide low magnitude and high frequency vibration treatment, which is self-developed by our research team

INTERVENTIONS:
Procedure: vibration platform provide low magnitude and high frequency vibration treatment, which is self-developed by our research team — Stand on a vibration platform at 35Hz, 0.3g, 20mins/day and 5days/week
  Arms: Treatment

SUMMARY:
Diaphyseal long bone fractures are usually associated with high energy trauma in which femoral shaft fracture is one common fracture in young age group. Surgery is usually needed for the diaphyseal lone bone fractures and the painful conditions always hinder weight bearing which is important for fracture healing and functional recovery. Fracture healing in cortical bone is less predictable than trabecular bone because they are less active and blood supply is more critical. Therefore accelerating fracture healing and rehabilitation of long bone fracture will absolutely bring significant economic benefit to the society in term of hospitalization and sick leave cost.

Low-magnitude, high-frequency vibration (LMHFV) treatment can provide systemic mechanical stimulation and is reported with multiple effects on musculoskeletal tissues. LMHFV can enhance the blood circulation and osteogenic effect in normal subjects and animals. Our previous clinical study also indicated that LMHFV could enhance the balancing ability and muscular function in normal post-menopausal women after treating whole-body vibration. For the fracture healing effect, an acceleration of healing by inducing callus formation and maturation in rat model was also reported in our previous studies.

In this study a total of 50 unilateral closed femoral shaft fracture patients of either gender aged 20-40 years old will be recruited and they will be randomized to either control and vibration group. The vibration group will be treated with LMHFV for 6 months. The findings of this study will provide very useful scientific data to support the application of LMHFV for fracture healing.

ELIGIBILITY:
Inclusion Criteria:

* male or non-pregnant female aged 20-40 years old
* patient with unilateral femoral shaft fracture
* Fractures fixed with titanium intramedullary nail
* patient able to comply with study protocol including follow evaluation

Exclusion Criteria:

* open fracture
* bilateral fracture
* patient with multiple system injuries
* fracture gap > 10mm
* pathologic fracture
* pregnant women
* history of medication or disease affecting bone metabolism such as hypo- or hyperparathyroidism and hypo-, hyperthyroidism

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time to radiologic healing | 1 year
  The healing time of fracture site among subjects is assessed by noting the time of appearance of the first bridging callus in x-ray film as well as the second bridging callus and the third bridging callus

SECONDARY OUTCOMES:
Functional outcomes | 1 year
  The subjects are needed to perform functional outcome measurement according to our established protocol, including quality of life, muscle strength, balancing ability, vertical jump performance. The result of the above assessments will be reported as a scoring to show the functional performance and mobility of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Kwok Sui Leung, MD, Principal Investigator — Department of Orthopaedics and Traumatology, The Chinese University of Hong Kong
Locations (1):
- Department of Orthopaedics and Traumatology , The Chinese University of Hong Kong, Hong Kong, China